CLINICAL TRIAL: NCT04225143
Title: Efficacité Clinique comparée de la Stimulation transcutanée du Nerf Tibial postérieur unilatérale vs bilatérale Pour Traiter Une hyperactivité vésicale Neurologique Non sévère : Essai Clinique randomisé
Brief Title: Bilateral vs. Unilateral Stimulation in Neurological Bladder Disroders
Acronym: UROSTIM
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Caen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UROSTIM
Record Dates: First submitted 2019-12-12; First posted 2020-01-13 (Actual); Last update posted 2020-01-13 (Actual); Status verified 2019-11

CONDITIONS: Neurogenic Urinary Bladder, Spastic
MeSH Terms: conditions — Urinary Bladder, Neurogenic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- bilateral (Experimental): 25 patients with an overactive bladder
  Interventions: Procedure: urostim bilateral
- unilateral (Active Comparator): 25 patients with an overactive bladder
  Interventions: Procedure: urostim unilateral

INTERVENTIONS:
Procedure: urostim bilateral — Treatment by bilateral neurostimulation of the tibial nerve
  Arms: bilateral
Procedure: urostim unilateral — Treatment by unilateral neurostimulation of the tibial nerve
  Arms: unilateral

SUMMARY:
This study evaluates the effectiveness of bilateral stimulation of the tibial nerve compared to unilateral stimulation in neurological bladder disorders.

DETAILED DESCRIPTION:
Urinary disorders are common in neurological diseases. The prognosis of neurological bladders is twofold. On the one hand, symptoms such as incontinence or retention affect quality of life and comfort. On the other hand, complications such as urinary tract infections or renal failure threaten health and even involve patients' vital prognosis. Several therapies are used to treat these urinary disorders including transcutaneous or percutaneous posterior tibial nerve stimulation (SNTP). SNTP is used in treating symptoms of bladder overactivity. This treatment is most often used unilaterally, but can be used bilaterally.

The aim of this study is to evaluate the effectiveness of bilateral stimulation of the tibial nerve compared to unilateral stimulation in neurological bladder disorders.

50 patients will be included, in two arms by randomization, one arm of 25 patients will be treated by unilateral stimuylation and the other arm of 25 patients will be trated by bilateral stimulation.

They will be evaluate at 3, 6 and 12 months by auto questionnaire and the effectivess of each therapy will be compared.

ELIGIBILITY:
Inclusion Criteria:

* Individuals who received research information
* Individuals affiliated to a social security scheme
* Individuals over 18 years of age
* Individuals with non-serious neurological bladder hyperactivity

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2019-11-27 (Actual); Primary Completion 2020-10-31 (Estimated); Study Completion 2021-10-31 (Estimated)

PRIMARY OUTCOMES:
Urinary symptom profile score (USP score) | 3 months
  auto quastionnaire between 0 and 39 points The higher the score the higher the urinary symptoms

SECONDARY OUTCOMES:
mictional calendar | 3 months
  records the number of mictions per day and the number of urinary leaks per day over 48 hours
Patient global impression of improvement (PGI-I) | 3 months
  Questionnaire of quality of life improvement :The PGI-I is a transition scale that is a single question asking the patient to rate their urinary tract condition now, as compared with how it was prior to before beginning treatment on a scale from 1 (Very much better) to 7 (Very much worse)

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Caen Normandie, Caen, France

IPD SHARING:
Plan to Share IPD: No